CLINICAL TRIAL: NCT07166237
Title: Group Cognitive Behavioural Therapy for Paternal Perinatal Depression: A Pilot Randomized Controlled Trial
Brief Title: Group Cognitive Behavioural Therapy for Paternal Perinatal Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBT for Paternal PND Pilot RCT
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Perinatal Depression; Fathers
Keywords: cognitive behavioral therapy; paternal depression; perinatal depression; fathers
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A parallel-group Ontario-wide RCT with experimental (9-week CBT + TAU) and control (TAU) groups will address our objectives. Participants will be randomly assigned in a 1:1 ratio to the treatment or control groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and the research coordinator cannot be blinded to group condition though the research assistants making reminder calls and data analysts will not be aware of group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9-Week Group Cognitive Behavioural Therapy Intervention (Experimental): The experimental group will receive a 9-week group CBT intervention delivered by a psychiatrist and a public health nurse in addition to receiving treatment as usual.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Paternal Perinatal Depression
- Control/Usual Care (No Intervention): Participants randomized to the No Intervention group will continue to receive treatment as usual (standard care). A list of resources will be emailed.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Paternal Perinatal Depression — Cognitive Behavioral Therapy (CBT) is a type of psychotherapy (talk therapy). The weekly group sessions will be two hours long and take place once a week for 9 consecutive weeks. The first hour of the session will involve teaching and practice of CBT skills, followed by one hour of unstructured discussion around topics relevant to participants with paternal perinatal depression. Each group will be delivered online via Zoom and guided by our intervention manual.
  Arms: 9-Week Group Cognitive Behavioural Therapy Intervention

SUMMARY:
The purpose of this pilot randomized controlled trial is to assess the feasibility of offering a 9-week group cognitive behavioural therapy (CBT; a type of talking therapy) led by a psychiatrist and public health nurse to fathers and non-birthing parents who identify as fathers or fathers-to-be (have a partner who is expecting) with perinatal depression. Fathers or fathers-to-be living in Ontario who have depression symptoms while their partner has been pregnant and/or during the first 18 months of their child's life will be assigned with a 50/50 chance (like flipping a coin) to receive online group CBT in addition to usual care, or to receive usual care only.

DETAILED DESCRIPTION:
This study will involve a pilot randomized controlled trial (RCT) to determine the feasibility of the intervention and study protocol for assessing if a 9-week group CBT intervention added to treatment as usual (TAU) can improve paternal perinatal depression symptoms more than TAU alone. The primary objective is to assess feasibility of the intervention including recruitment, completion of study measures, retention, and participant satisfaction/acceptability of the intervention. The secondary objective of the RCT is to estimate treatment effects on depressive symptoms to guide the conduct of a future full-scale RCT of the intervention. Estimate of treatment effect will serve as a primary outcome measure in a later full-scale RCT.

Forty-eight participants will be assigned in a 1:1 ratio to the experimental or control group. Participants in both groups will complete online questionnaires and structured telephone interviews at baseline (T1), 9 weeks later (T2 - immediately post-intervention in the experimental group) and 6 months post-enrollment (T3). Those assigned to receive the 9-week CBT group will also be asked questions about their satisfaction with the program and recommendations for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Non-birthing individuals identifying as fathers-to-be (i.e., have a pregnant partner) or fathers with an infant <18 months at recruitment, be fluent in written/spoken English, have an EPDS score ≥9 and live in Ontario

Exclusion Criteria:

* Free of bipolar, psychotic, borderline personality and current substance use disorders

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited in recruitment period | 6 months
  Recruit and randomize 48 participants (over two groups; 24 experimental, 24 control) in six months
Number of participants who complete all data collection procedures | 6 months
  75% of participants complete all three questionnaires and structured interviews
Number of participants who complete study (retention) | 6 months
  75% of participants remain in study until completion
Number of participants who complete the intervention (adherence) | 6 months
  80% of participants in treatment group complete the intervention

SECONDARY OUTCOMES:
Estimate treatment effect - Edinburgh Postnatal Depression Scale (EPDS) | 9 weeks
  Perinatal depression (PND) is best conceptualized as a continuous construct with its impact operating across a continuum of severity, and so a continuous measure of PND (EPDS) is our primary outcome. In keeping with most PND RCTs, our primary effectiveness time point is immediately post-treatment (T2). We will also assess the durability of intervention effects at three months post-T2 (T3). The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item gold standard measure of PND. Total scores range from 0-30 with higher scores indicating worse depressive symptoms. A score of ≥10 is consistent with possible PND, ≥13 is consistent with probable PND and changes in scores >4 are accepted as being indicative of clinically significant change.

OTHER OUTCOMES:
Estimate treatment effect - Edinburgh Postnatal Depression Scale (EPDS) | 6 months
  Perinatal depression (PND) is best conceptualized as a continuous construct with its impact operating across a continuum of severity, and so a continuous measure of PND (EPDS) is our primary outcome. In keeping with most PND RCTs, our primary effectiveness time point is immediately post-treatment (T2). We will also assess the durability of intervention effects at three months post-T2 (T3). The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item gold standard measure of PND. Total scores range from 0-30 with higher scores indicating worse depressive symptoms. A score of ≥10 is consistent with possible PND, ≥13 is consistent with probable PND and changes in scores >4 are accepted as being indicative of clinically significant change.
Major Depressive Disorder | 9 weeks
  A structured psychiatric interview will assess current psychiatric syndromes in participants. The Diagnostic Assessment Research Tool (DART) will be conducted at baseline, T2 and T3 to assess change in psychiatric symptoms over the study period.
Major Depressive Disorder Module | 6 months
  A structured psychiatric interview will assess current psychiatric syndromes in participants. The Diagnostic Assessment Research Tool (DART) will be conducted at baseline, T2 and T3 to assess change in psychiatric symptoms over the study period.
General Anxiety Disorder (GAD-7) | 9 weeks
  A reliable and valid 7-item self-report scale that assesses the symptoms of generalized anxiety disorder, the most common comorbidity of PND. A cutoff of ≥10 defines clinically important levels of anxiety symptoms and changes in scores >4 are accepted as being indicative of clinically significant change.
General Anxiety Disorder (GAD-7) | 6 months
  A reliable and valid 7-item self-report scale that assesses the symptoms of generalized anxiety disorder, the most common comorbidity of PND. A cutoff of ≥10 defines clinically important levels of anxiety symptoms and changes in scores >4 are accepted as being indicative of clinically significant change.
Parenting Stress Index - Short Form | 9 weeks
  The Parenting Stress Index (Short Form) is a 36-item parent self-report measure that identifies potentially dysfunctional parent-child systems on three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. The measure also produces a total score that is an indication of overall level of stress a person is feeling in their role as a parent. Higher scores indicate higher levels of stress.
Parenting Stress Index - Short Form | 6 months
  The Parenting Stress Index (Short Form) is a 36-item parent self-report measure that identifies potentially dysfunctional parent-child systems on three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. The measure also produces a total score that is an indication of overall level of stress a person is feeling in their role as a parent. Higher scores indicate higher levels of stress.
Multidimensional Scale of Perceived Social Support (MSPSS) | 9 weeks
  A 12-item scale designed to measure perceived social support from three sources: (1) family, (2) friends and (3) significant other. Items are scored on a 7-point scale, and total scores range from 12-84 with higher scores indicating a higher level of perceived social support. A score of 12-35 indicates low perceived social support, 36-60 indicates medium perceived social support and 61-84 indicates high perceived social support.
Multidimensional Scale of Perceived Social Support (MSPSS) | 6 months
  A 12-item scale designed to measure perceived social support from three sources: (1) family, (2) friends and (3) significant other. Items are scored on a 7-point scale, and total scores range from 12-84 with higher scores indicating a higher level of perceived social support. A score of 12-35 indicates low perceived social support, 36-60 indicates medium perceived social support and 61-84 indicates high perceived social support.
Dyadic Adjustment Scale (DAS) | 9 weeks
  The Dyadic Adjustment Scale (DAS) will be used to measure an individual's feelings about their relationship with an intimate partner. The scale contains 32-item with items scored on 2-, 5-,6-, or 7-point scales. The DAS contains four subscales: dyadic consensus, dyadic satisfaction, dyadic cohesion, and affective expression. Total scale scores were used in this study, with higher scores indicating greater relationship satisfaction.
Dyadic Adjustment Scale (DAS) | 6 months
  The Dyadic Adjustment Scale (DAS) will be used to measure an individual's feelings about their relationship with an intimate partner. The scale contains 32-item with items scored on 2-, 5-,6-, or 7-point scales. The DAS contains four subscales: dyadic consensus, dyadic satisfaction, dyadic cohesion, and affective expression. Total scale scores were used in this study, with higher scores indicating greater relationship satisfaction.
Postpartum Bonding Questionnaire (PBQ) | 9 weeks
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item parent-report measure that assesses four aspects of father-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Father-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Postpartum Bonding Questionnaire (PBQ) | 6 months
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item parent-report measure that assesses four aspects of father-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Father-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Infant Behavior Questionnaire-Revised Very Short Form (IBQ-R VSF) | 9 weeks
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
Infant Behavior Questionnaire-Revised Very Short Form (IBQ-R VSF) | 6 months
  The Infant Behaviour Questionnaire-Revised (Very Short Form) (IBQR) is a parent-report measure of infant temperament. The IBQ-R (Very Short Form) consists of 37 items answered on a 7-point scale (1-7) and assesses 3 factors: Positive Affectivity/Surgency with 13 items, Negative Emotionality with 12 items, and Orienting/Regulatory Capacity with 12 items; higher scores indicate greater alignment with the domain.
Maternal Perinatal Depression - Edinburgh Postnatal Depression Scale (EPDS) | 9 weeks
  To assess maternal perinatal depression (PND), partners of fathers participating in the study will complete the EPDS. The EPDS is a 10-item gold standard measure of PND. Total scores range from 0-30 with higher scores indicating worse depressive symptoms. A score of ≥10 is consistent with possible PND, ≥13 is consistent with probable PND and changes in scores >4 are accepted as being indicative of clinically significant change.
Maternal Perinatal Depression - Edinburgh Postnatal Depression Scale (EPDS) | 6 months
  To assess maternal perinatal depression (PND), partners of fathers participating in the study will complete the EPDS. The EPDS is a 10-item gold standard measure of PND. Total scores range from 0-30 with higher scores indicating worse depressive symptoms. A score of ≥10 is consistent with possible PND, ≥13 is consistent with probable PND and changes in scores >4 are accepted as being indicative of clinically significant change.
Healthcare Resource Utilization | 9 weeks
  Healthcare resource utilization data will be collected using a questionnaire used in prior work and adapted for the postpartum period (based on the Canadian Community Health Survey and Service Use and Resources Form). Participants will provide information on all healthcare service and medication use from T1 to T3 from the perspective of the public health care payer.
Healthcare Resource Utilization | 6 months
  Healthcare resource utilization data will be collected using a questionnaire used in prior work and adapted for the postpartum period (based on the Canadian Community Health Survey and Service Use and Resources Form). Participants will provide information on all healthcare service and medication use from T1 to T3 from the perspective of the public health care payer.
Quality-Adjusted Life Year (QALY) | 9 weeks
  The EQ-5D-5L is a utility-based health-related quality of life instrument assessing five domains (mobility, self-care, usual activities, pain, depression/anxiety) and will be administered at T1-T3. Its validity in measuring the impact of depression is established. We will use its Canadian algorithm to convert responses to health utility. QALYs will be calculated by multiplying the health utility for the corresponding time period (i.e., area under the curve approach).
Quality-Adjusted Life Year (QALY) | 6 months
  The EQ-5D-5L is a utility-based health-related quality of life instrument assessing five domains (mobility, self-care, usual activities, pain, depression/anxiety) and will be administered at T1-T3. Its validity in measuring the impact of depression is established. We will use its Canadian algorithm to convert responses to health utility. QALYs will be calculated by multiplying the health utility for the corresponding time period (i.e., area under the curve approach).
Client Satisfaction Questionnaire (CSQ-8) | 9 weeks
  Intervention participants only. We will assess participant satisfaction with the intervention using the eight-item Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 consists of eight items assessing the level of satisfaction with the intervention on a 4-point Likert-type scale, as well as one open-ended question. Responses to the open-ended question will be analyzed using content analysis to inform acceptability of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No